CLINICAL TRIAL: NCT05530395
Title: Baseline Testosterone as a Prognostic and/or Predictive Biomarker in Metastatic Hormone Sensitive Prostate Cancer
Brief Title: BAseLine TEstosterone as a Prognostic and/or Predictive bioMARKer in mHSPC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ignacio Puche Sanz (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitario Torrecárdenas (Other); Hospital Neurotraumatologico de Jaen (Other); Hospital San Carlos, Madrid (Other); Institut Mutualiste Montsouris (Other); San Raffaele University Hospital, Italy (Other); Azienda Ospedaliera San Giovanni Battista (Other); Chinese University of Hong Kong (Other); Medical University Innsbruck (Other); University of Padova (Other); UMC Utrecht (Other)
Responsible Party: Sponsor-Investigator, Ignacio Puche Sanz, Principal Investigator, University Hospital Virgen de las Nieves
Organization: University Hospital Virgen de las Nieves (Other)
Other Study IDs: BATEMARK-YAUPCa-21
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer Metastatic
Keywords: Testosterone, biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Testosterone levels — Blood sample to determine testosterone levels

SUMMARY:
Despite large amounts of basic-science data supporting a role for androgens in PCa pathogenesis, there are conflicting clinical data on the role of endogenous testosterone in human de novo PCa pathogenesis. The investigators hypothesize that lower baseline serum testosterone is significantly associated with worse clinical outcomes in mHSPC patients undergoing continuous medical castration

DETAILED DESCRIPTION:
Biological rationale:

The 'androgen hypothesis' asserts that prostate cancer (PCa) development and progression is driven by androgens. There is significant evidence that androgens promote prostate cancer in experimental models. However, there is no clear evidence that elevations in endogenous testosterone levels promote the development of prostate cancer in humans. Indeed, despite large amounts of basic-science data supporting a role for androgens in PCa pathogenesis, there are conflicting clinical data on the role of endogenous testosterone in human PCa pathogenesis de novo. In reviewing the literature involving PCa development in PCa naive patients, there are studies implicating elevated testosterone, studies implicating lower testosterone, and studies with no association of testosterone and PCa risk.

A recent review in 2015 delved into the controversial role of androgens and prostate cancer and explains the different theories about the ambiguous action of testosterone on the prostate. In 2012, a research proposed the nonlinear U-shaped behaviour or time dependency theory, which postulates that the endocrine biology of the prostate tissue depends on exposure time at a given androgen concentration, which "relies on the fluctuation of the levels of circulating sex steroids during the lifespan of the individual". Another model is the saturation model based on the observations that prostate tissue is extremely sensitive to changes in serum testosterone at low concentrations. This model suggests that there is a nonprotective effect of low testosterone against PCa but tissue becomes indifferent to changes when increasing androgen concentration reach a limit (saturation point), beyond which no further androgen-driven changes are observed. Anyway, the lack of a satisfying model to explain the relationship between androgens and PCa is simply the consequence of insufficient knowledge of the real intrinsic physiopathology of this disease.

Clinical rationale:

Approximately 15% of mHSPC patients primarily fail to respond to ADT. A recent consensus statement on circulating biomarkers for advanced prostate cancer highlighted the urgent need for prospective trials to clinically qualify circulating biomarkers, the greatest need being metastatic PCa. On the other hand, a very recent paper analysed baseline testosterone in hormone-naïve advanced PCa patients undergoing continuous medical castration and selected from 2 large Phase III RCTs. It demonstrated that lower baseline serum testosterone was significantly associated with worse survival end-points and warrants further prospective research in this scenario.

In this era of complex and expensive next-generation markers, this simple, cheap, and well-known biomarker may still have something to say in PCa.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic hormone sensitive prostate cancer (mHSPC) patients diagnosed by any imaging test (at least CT and bone scan) including:

  * Any newly diagnosed mHSPC with no prior treatments.
  * Primarily treated PCa that have progressed to mHSPC with no prior ADT in the last 2 years.
  * Patients receiving ADT + EBRT as primary treatment will also be included.
* Patients who agree to be followed prospectively according to routine clinical practice in the context of this study.

Exclusion Criteria:

* Any prior androgen deprivation therapy (ADT) scheme 2 years before recruitment. - Any prior testosterone replacement therapy scheme 2 years before recruitment.
* Previous intermittent ADT schemes.
* Prior testicular excision surgery.
* Absence or testicular atrophy from any cause.
* Whenever further prospective clinical follow-up is not possible or patient do not accept follow-up in the context of this study.

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic hormone sensitive prostate cancer (mHSPC) patients diagnosed by any imaging test (at least CT and/or bone scan).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Early treatment failure | 1 year
  Proportion of patients with PSA progression or death from PCa within 12 months after initiation of treatment.
PSA response | 6 months
  Lowest PSA (nadir) reached after initiation of treatment

SECONDARY OUTCOMES:
Testosterone response. | 6 months
  %percent of decrease in testosterone levels at the moment of PSA nadir.
Biochemical progression-free survival (bPFS) | 1 year
  PSA progression: 2 consecutive increase at least 50% or 5 ng/mL or more above PSA nadir on 2 consecutive measurements at least 2 weeks apart.
Radiologic progression-free survival (rPFS) | 1 year
  Assessed by PCWG3 progression criteria on nodal, visceral and bone disease.
Time to CRPC | 1 year
  Time (months) from treatment initiation to the development of a CRPC status.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Puche, Principal Investigator — Fundación para la Investigación Biosanitaria de Andalucía Oriental (FIBAO)
Locations (3):
- Spain (3):
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michaud JE, Billups KL, Partin AW. Testosterone and prostate cancer: an evidence-based review of pathogenesis and oncologic risk. Ther Adv Urol. 2015 Dec;7(6):378-87. doi: 10.1177/1756287215597633. PMID 26622322
- [Background] Pierorazio PM, Ferrucci L, Kettermann A, Longo DL, Metter EJ, Carter HB. Serum testosterone is associated with aggressive prostate cancer in older men: results from the Baltimore Longitudinal Study of Aging. BJU Int. 2010 Mar;105(6):824-9. doi: 10.1111/j.1464-410X.2009.08853.x. Epub 2009 Sep 14. PMID 19751256
- [Background] Yano M, Imamoto T, Suzuki H, Fukasawa S, Kojima S, Komiya A, Naya Y, Ichikawa T. The clinical potential of pretreatment serum testosterone level to improve the efficiency of prostate cancer screening. Eur Urol. 2007 Feb;51(2):375-80. doi: 10.1016/j.eururo.2006.08.047. Epub 2006 Sep 12. PMID 17005316
- [Background] Rajek NJ. Developing an evening clinical experience for baccalaureate community health nursing students. J Nurs Educ. 1987 May;26(5):197-200. doi: 10.3928/0148-4834-19870501-07. PMID 3035140